CLINICAL TRIAL: NCT03544411
Title: Effects of Olive Oil and Bran Oil on Antioxidant Levels, Glycemic Control, and Lipid Profile in Patient Diabetes Mellitus Type 2
Brief Title: Effects of Olive Oil and Bran Oil on Antioxidant Levels, Glycemic Control, and Lipid Profile in Patient Type 2 DM
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Indonesia University (Other)
Collaborators: Fakultas Kedokteran Universitas Indonesia (Other)
Responsible Party: Principal Investigator, Rina Agustina, Head of Human Nutrition Research Centre, Indonesia University
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BeZaproject
Record Dates: First submitted 2018-05-19; First posted 2018-06-01 (Actual); Last update posted 2018-10-16 (Actual); Status verified 2018-10

CONDITIONS: Diabetes Mellitus, Type 2; Oxidative Stress; Glucose, High Blood; Lipid Disorder
Keywords: Olive oil; Bran oil; Type 2 Diabetes Mellitus; Antioxidant; glycemic control; lipid profile
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Lipid Metabolism Disorders | interventions — Olive Oil; Rice Bran Oil

STUDY DESIGN:
Intervention Model Description: This study was a clinical trial with cross over study design, random allocation, and double blindness to compare changes in antioxidant, glucose, cholesterol and triglyceride levels supplemented with 15 ml / day of olive oil (KZ) with supplementation of 15 ml / day of bran oil (KB). Provision of oil for 4 weeks in a row. During the 2-week interval not being treated (wash out). After the wash out period cross-over by exchanging olive oil supplementation to rice bran and vice versa for 4 consecutive weeks.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Type 2 Diabetes Mellitus group 1 (Experimental): The group supplemented with 15 ml / day of olive oil and 15 ml / day of bran oil
  Interventions: Biological: olive oil; Biological: bran oil
- Type 2 Diabetes Mellitus group 2 (Experimental): this group supplemented with 15 ml / day of olive oil and 15 ml / day of bran oil
  Interventions: Biological: olive oil; Biological: bran oil

INTERVENTIONS:
Biological: olive oil — the intervention consist of 15 ml / day of olive oil
Biological: bran oil — the intervention consist of 15 ml / day of bran oil

SUMMARY:
This study determines the effect of olive oil and bran oil on antioxidant levels, and glycemic control in patients with type 2 diabetes mellitus (DM)

Intervention: Patient type 2 DM will receive olive oil and bran oil with cross over study

DETAILED DESCRIPTION:
Diabetes mellitus (DM) has become one of the global public health problems. The chronic complications of type 2 DM can be macrovascular and microvascular complications that can decrease the quality of life of the patient. The main goal of sustainable DM nutrition therapy is to keep glucose in the blood close to normal levels to stop hyperglycemic and hyperlipidemic events that may inhibit further complications

This study was a clinical trial with cross over study design, random allocation, and double blindness to compare changes in antioxidant, glucose, cholesterol and triglyceride levels supplemented with 15 ml / day of olive oil (KZ) with supplementation of 15 ml / day of bran oil (KB). Provision of oil for 4 weeks in a row. During the 2-week interval not being treated (wash out). After the wash out period cross-over by exchanging olive oil supplementation to rice bran and vice versa for 4 consecutive weeks. The research will be conducted at Family Clinic Clinic FKUI Kayu Putih, Jakarta.

ELIGIBILITY:
Inclusion Criteria:

* Patients with type 2 diabetes aged 30-60 years.
* Diagnosed type 2 DM <3 years.
* Body mass index of 20-30 kg / m2
* Subjects willing to participate in research and sign informed consent.
* Drinking OHO (oral hyperglycemic medication).

Exclusion Criteria:

* There are acute and chronic complications.
* Subject is pregnant.
* Get cholesterol-lowering drugs, steroids and other drugs that affect the metabolism of fat.
* Smoking more than 10 cigarettes / day.
* Eat regular supplements that contain phytosterols or other antioxidants that are known by anamnesis.
* Has a disorder or gastrointestinal disease, thyroid, heart, liver, cancer, stroke and kidney are known with medical record data.

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2018-07-02 (Actual); Primary Completion 2018-09-20 (Actual); Study Completion 2018-10-05 (Actual)

PRIMARY OUTCOMES:
Change of malondialdehyde | baseline at Day0 and ,midline at Day28 and endline at Day70
  Change from baseline malondialdehyde at 4 weeks and at 10 weeks, is measured in pmol/mL

SECONDARY OUTCOMES:
Change of fasting plasma glucose | baseline at Day0 and ,midline at Day28 and endline at Day70
  Change from baseline fasting plasma glucose at 4 weeks and at 10 weeks, is measured in mg/dL
Change of post prandial blood glucose | baseline at Day0 and ,midline at Day28 and endline at Day70
  Change from baseline post prandial blood glucose at 4 weeks and at 10 weeks, is measured in mg/dL
Change of total cholesterol | baseline at Day0 and ,midline at Day28 and endline at Day70
  Change from baseline cholesterol at 4 weeks and at 10 weeks, is measured in mg/dL
Change of Low density lipoprotein | baseline at Day0 and ,midline at Day28 and endline at Day70
  Change from baseline Low density lipoprotein at 4 weeks and at 10 weeks, is measured in mg/dL
Change of High density lipoprotein | baseline at Day0 and ,midline at Day28 and endline at Day70
  Change from baseline High density lipoprotein at 4 weeks and at 10 weeks, is measured in mg/dL
Change of Trygliseride | baseline at Day0 and ,midline at Day28 and endline at Day70
  Change from baseline trygliseride at 4 weeks and at 10 weeks, is measured in mg/dL
Change of Katalase | baseline at Day0 and ,midline at Day28 and endline at Day70
  Change from baseline katalase at 4 weeks and at 10 weeks, is measured in unit/ mg protein
Change of Superoxide Dismutase | baseline at Day0 and ,midline at Day28 and endline at Day70
  Change from baseline superoxide dismutase at 4 weeks and at 10 weeks, is measured in unit/ mg protein
Change of Glutahione | baseline at Day0 and ,midline at Day28 and endline at Day70
  Change from baseline gluthatione at 4 weeks and at 10 weeks, is measured in nmol/ gram

CONTACTS AND LOCATIONS:
Overall Officials: Dwirini R Gunarti, DR, Principal Investigator — Indonesia University
Locations (1):
- Fkui-Kdk Kiara, Jakarta Pusat, DKI Jakarta, Indonesia